CLINICAL TRIAL: NCT04321746
Title: The Effect of Ketamine on Postoperative Cognitive Dysfunction in Geriatric Patients Undergoing Orthopaedic Surgery Under Spinal Anaesthesia, a Randomized Controlled Trial
Brief Title: The Effect of Ketamine on Postoperative Cognitive Dysfunction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ketamine
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Active Comparator)
  Interventions: Drug: Ketamine
- Control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — ketamine will be administered at a dose of 0.3 mg/kg in normal saline at 0.9% (250 mL)
  Arms: Ketamine
Other: Placebo — the control group will receive only normal saline at 0.9%, with the same physical characteristics of the ketamine solution
  Arms: Control

SUMMARY:
Available evidence suggests that there is no significant difference in the incidence of postoperative cognitive dysfunction POCD when general anaesthesia and regional anaesthesia are compared[13, 14]. To the knowledge of the investigators , no studies are examining the effects of ketamine on cognitive outcomes in the setting of spinal anesthesia.

Thus, the purpose of this study was to compare the cognitive status, as assessed by the SPMSQ, of elderly patients undergoing orthopaedic surgery under spinal anaesthesia before and after ketamine administration. The authors hypothesized that patients receiving ketamine would exhibit better cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for orthopaedic surgery under spinal anaesthesia.
* ASA physical status I to II.

Exclusion Criteria:

* Patients with a history of psychosis, schizophrenia, nephropathy, uncontrolled blood pressure, uncontrolled hepatic disorders, or allergy to ketamine.
* Patients With moderate to severe depression according to Yesavage abbreviated Geriatric Depression Scale,
* Patients presented with postoperative delirium or required medications other than study drugs.
* Ketamine administration is contraindicated.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
postoperative cognitive dysfunction | first postoperative day
  cognitive status will be conducted with the Short Portable Mental Status Questionnaire SPMSQ preoperative and 2 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No